CLINICAL TRIAL: NCT03827239
Title: Investigation of the Effects of Sedentary Behaviour and Moderate Exercise on Glucose Tolerance and Insulin Sensitivity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding caused us to cancel the study.
Sponsor: University of Prince Edward Island (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 6007895
Record Dates: First submitted 2019-01-22; First posted 2019-02-01 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2019-01

CONDITIONS: Sedentary Lifestyle; Insulin Sensitivity; Glucose Metabolism
MeSH Terms: conditions — Sedentary Behavior; Insulin Resistance | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No intervention. Study participants will be seated during the entire sedentary 3-hour time period and wheeled to phlebotomy (and exercise) stations when required. During the sedentary period, participants will eat the food according to the study protocol and be seated at desks and allowed to read and use computers.
- Intervention (Experimental): Will disrupt their sedentary time with 3 minute exercise sessions every 30 minutes
  Interventions: Other: Activity/Moderate Exercise

INTERVENTIONS:
Other: Activity/Moderate Exercise — 3-hour sedentary period with 3 minute activity breaks of moderate exercise every 30 minutes
  Arms: Intervention

SUMMARY:
Individuals with pre-diabetes or diabetes would benefit from low impact methods that would improve their insulin sensitivity and aid in maintaining glucose homeostasis. Physical activity helps the body decrease its insulin resistance and burn excess sugar. Many diabetics also suffer from obesity and specific forms or durations of physical exercise may not be viable options for these individuals. Determining whether short bursts of moderate exercise improve blood glucose levels in healthy humans may identify a further method for diabetics to improve their glucose homeostasis.

The aim of this study is to determine the most effective moderate exercise that can be completed in 3 minutes and its effectiveness on improving glucose handling, in response to a single day of standardized high-fat and high-carbohydrate feeding in comparison to periods of prolonged sitting.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* BMI between 18-30 kg/m²
* non-smoker

Exclusion Criteria:

* pregnant
* diabetes
* kidney disease
* liver disease
* cardiovascular disease
* cancer

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Insulin levels | Pre-prandial baseline (12 hours fasted) and 3 hours post-prandial on each of two testing days
  The change in blood insulin levels from baseline (12 hours fasted) to 3-hours post-prandial will be determined from blood serum using a human metabolic hormone multiplex panel (Luminex xMAP technology).
Change in concentration of C-peptide | Pre-prandial baseline (12 hours fasted) and 3 hours post-prandial on each of two testing days
  The change in blood C-peptide levels from baseline (12 hours fasted) to 3-hours post-prandial will be determined from blood serum using a human metabolic hormone multiplex panel (Luminex xMAP technology).
Changes in blood glucose levels | Baseline and every 30-60 minutes over 3 hours (6 timepoints per test day)
  Blood glucose levels will be determined at pre-prandial baseline and over the following 3-hour testing period using hand-held blood glucose meters.
Change in metabolomic response to a test meal | Pre-prandial and 3-hours post test meal through study completion
  Targeted metabolomics analysis of approximately 139 metabolites in blood serum by LC-MS/MS to generate a metabolomic profile in response to a high-fat and high-carbohydrate test meal. Metabolites to be determined are categorized as biogenic amines, amino acids, histidines, carboxylic acids, acylcarnitines, glycerophospholipids and organic acids.

SECONDARY OUTCOMES:
Immediate effects of short-term sedentary behaviour on cognitive function | 3 hours post-activity (sedentary behaviour or exercise) on test days through study completion
  Assessing cognitive abilities using the Stroop Test.
Immediate effects of short-term sedentary behaviour on cognitive function | 3 hours post-activity (sedentary behaviour or exercise) on test days through study completion
  Assessing cognitive abilities using the Iowa Trail Making Test.
Immediate effects of short-term sedentary behaviour on cognitive function | 3 hours post-activity (sedentary behaviour or exercise) on test days through study completion
  Assessing cognitive abilities using the Digit-Span test.
Immediate effects of short-term sedentary behaviour on cognitive function | 3 hours post-activity (sedentary behaviour or exercise) on test days through study completion
  Assessing cognitive abilities using the N-back test.
Immediate effects of short-term sedentary behaviour on cognitive function | 3 hours post-activity (sedentary behaviour or exercise) on test days through study completion
  Assessing cognitive abilities using the Flankers test.
Gene expression levels in isolated PBMC populations | Pre-prandial and 3 hours post-prandial on on test days through study completion
  Determining changes in gene expression in pathways associated with RAGE signalling.

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Mahlstedt, PhD, Study Director — University of Prince Edward Island
Locations (1):
- University of Prince Edward Island, Charlottetown, Prince Edward Island, Canada